CLINICAL TRIAL: NCT00005991
Title: Phase I/II Study of Gemcitabine and Doxil Combination Chemotherapy in Patients With Advanced Solid Tumors (Phase I)/Breast Cancer (Phase II)
Brief Title: Gemcitabine and Liposomal Doxorubicin in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067980; MDA-DM-97127; NCI-1650; DM97-127 (Other: UT MD Anderson Cancer Center)
Record Dates: First submitted 2000-07-05; First posted 2004-02-25 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: pegylated liposomal doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of gemcitabine and liposomal doxorubicin in treating women who have metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the objective response rate, duration of response, time to disease progression, and duration of survival of women with metastatic breast cancer when treated with gemcitabine and doxorubicin HCl liposome.

II. Determine the qualitative and quantitative toxicity and reversibility of toxicity of this treatment regimen in these patients.

OUTLINE: Patients receive gemcitabine intravenous (IV) over 30 minutes on days 1 and 8 and doxorubicin HCl liposome IV over 2.5 hours on day 1. Treatment continues every 21 days in the absence of disease progression or unacceptable toxicity. Patients are followed at 3 weeks.

PROJECTED ACCRUAL: A total of 22-46 patients will be accrued for this study within 20 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic breast cancer Bidimensionally measurable disease No uncontrolled brain metastases or leptomeningeal disease Brain metastases treated with surgery and/or radiotherapy allowed if neurologic status is stable two weeks after last dose of dexamethasone Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Sex: Female Menopausal status: Not specified Performance status: Zubrod 0-2 Life expectancy: At least 3 months Hematopoietic: Platelet count at least 100,000/mm3 Hemoglobin at least 8 g/dL Absolute neutrophil count at least 1,500/mm3 Hepatic: Bilirubin no greater than 1.2 mg/dL SGPT less than 1.5 times upper limit of normal Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: LVEF at least 50% by MUGA No cardiac disease or congestive heart failure Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No other concurrent serious illness, psychiatric disorder, or active infection No other prior or concurrent malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior high-dose chemotherapy followed by bone marrow transplantation Chemotherapy: See Biologic Therapy At least 3 weeks since prior chemotherapy and recovered No prior doxorubicin HCl liposome or gemcitabine Prior neoadjuvant chemotherapy allowed At least 12 months since prior adjuvant anthracycline-based therapy and no evidence of anthracycline resistance (i.e., developed progressive disease while receiving adjuvant therapy or within 6 months of completing adjuvant therapy) Prior mitoxantrone allowed if total dose was no greater than 105 mg/m2 IV bolus or 140 mg/m2 IV continuous infusion Prior doxorubicin allowed if total dose was no greater than 300 mg/m2 IV bolus or 400 mg/m2 IV continuous infusion No prior chemotherapy for metastatic disease Endocrine therapy: Prior adjuvant and/or palliative hormonal therapy allowed Radiotherapy: See Disease Characteristics At least 3 weeks since prior radiotherapy and recovered Surgery: See Disease Characteristics Prior surgery allowed Other: At least 3 weeks since prior investigational study Concurrent pamidronate allowed if bone not the only site of disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 1997-08-25 (Actual); Primary Completion 2003-02-14 (Actual); Study Completion 2003-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edgardo Rivera, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Background] Rivera E, Valero V, Esteva FJ, Syrewicz L, Cristofanilli M, Rahman Z, Booser DJ, Hortobagyi GN. Lack of activity of stealth liposomal doxorubicin in the treatment of patients with anthracycline-resistant breast cancer. Cancer Chemother Pharmacol. 2002 Apr;49(4):299-302. doi: 10.1007/s00280-001-0405-3. Epub 2001 Dec 18. PMID 11914909
- [Result] Rivera E, Valero V, Arun B, Royce M, Adinin R, Hoelzer K, Walters R, Wade JL 3rd, Pusztai L, Hortobagyi GN. Phase II study of pegylated liposomal doxorubicin in combination with gemcitabine in patients with metastatic breast cancer. J Clin Oncol. 2003 Sep 1;21(17):3249-54. doi: 10.1200/JCO.2003.03.111. PMID 12947059